CLINICAL TRIAL: NCT01331460
Title: HIV and Drug Use in Georgian Women
Acronym: IMEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA029880 (NIH); R01DA029880 (NIH)
Record Dates: First submitted 2011-02-22; First posted 2011-04-08 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; HIV risk; Sexually Transmitted Diseases; Drug Use; Women; Drug Treatment; opioids; injection drug use; stimulants; gender-specific treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Case Management

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RBT Experimental (Experimental)
  Interventions: Behavioral: RBT
- Case-Management: Treatment as Usual (Active Comparator)
  Interventions: Other: Case-Management

INTERVENTIONS:
Behavioral: RBT — Intervention for Injection Drug Using Women:
  Incorporates elements of Reinforcement-Based Treatment and Women's Health CoOp to help prevent drug abuse (and promote drug abstinence) and lower risk of Human Immunodeficiency Virus, violence, and high-risk sexual behaviors.
  Other Names: Women's Health CoOp
  Arms: RBT Experimental
Other: Case-Management — Standard Intervention:
  Incorporates standard practice elements like accessing resources, service linkage, monitoring the success of patient-service linkages, and advocating for the patient to help her meet her needs
  Other Names: Treatment-as-Usual; Standard Intervention
  Arms: Case-Management: Treatment as Usual

SUMMARY:
The purpose of this study is to determine how drug abuse treatment interventions can be integrated with established Human Immunodeficiency Virus prevention approaches to optimize their combined effectiveness.

DETAILED DESCRIPTION:
Eastern Europe is an emerging epicenter of injection drug use and Human Immunodeficiency Virus infection, among women. Within Eastern Europe, the Republic of Georgia is one of the last countries where an Human Immunodeficiency Virus epidemic can still be averted. This proposal responds to RFA-DA-10-008 International Research Collaborations on Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome and Drug Use by building on the successful collaboration among United States and Eastern European investigators from the Republic of Georgia and Russia. Recent data from Georgia's neighbor, Russia, reported 59% of Injection Drug Using women Human Immunodeficiency Virus seropositive; this is a threat that looms over Georgia. Understanding the risk factors that operate in Russia that drive this epidemic may help forestall such a catastrophe in Georgia. As such, this proposal directly responds to the Eastern European Region question of "How can drug abuse treatment interventions be integrated with established Human Immunodeficiency Virus prevention approaches to optimize their combined effectiveness?" Injection drug using Georgian women show prevalence rates of 2% for Human Immunodeficiency Virus and 25% for hepatitis C. The low prevalence of Human Immunodeficiency Virus in Georgian women provides an important window of opportunity to intervene and avoid the possibility of a Human Immunodeficiency Virus epidemic. In Georgia, women's expected subordination to men makes women vulnerable to Human Immunodeficiency Virus/Hepatitis C infection. The public health impact of the proposed project is far-reaching. Taken to scale, our Georgian reinforcement-based treatment model holds the promise not only to lessen the possibility of a Human Immunodeficiency Virus epidemic and slow the increase in the Hepatitis C transmission rate in Georgia, but also to strongly influence the development of women-focused drug abuse intervention models for treatment tailoring and dissemination in other nations.

ELIGIBILITY:
Inclusion Criteria:

* Conversant in Georgian
* Able to provide informed consent
* Age 18 years or older
* Has ever injected illicit drugs
* Sexually active at least once in the past 30 days.

Exclusion Criteria:

* Male
* Younger than 18 years
* Not sexually active at least once in past 30 days
* Not able to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-04; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sexual practices | 3 months after randomization
  Frequency of unprotected sexual acts in the past 30 days measured by revised risk behavior assessment
Injection Practices | 6 months after randomization
  Frequency of sharing other injection equipment in the past 30 days measured by revised risk behavior assessment
Injection practices | 3 months after randomization
  Frequency of sharing other injection equipment in the past 30 days measured by revised risk behavior assessment
Sexual Practices | 6 months after randomization
  Frequency of unprotected sexual acts in the past 30 days measured by revised risk behavior assessment

SECONDARY OUTCOMES:
Sexual practices | 3 months after randomization and 6 months after randomization
  Unprotected sex at last encounter measured by revised risk behavior assessment
Condom Use and Sexual Encounter Negotiation | 3 months after randomization and 6 months after randomization
  To use a condom in past 30 days and to negotiate sexual encounters in past 30 days measured by revised risk behavior assessment
Injecting practices | 3 months after randomization and 6 months after randomization
  Frequency of sharing other injection equipment in the past 30 days measured by revised risk behavior assessment
Drug use | 3 months after randomization and 6 months after randomization
  Frequency of opioid use in past 30 days revised risk behavior assessment plus urine test Self-Report verified by biological sample Poisson. Also frequency of stimulant use in past 30 days revised risk behavior assessment and urine test. Addiction Severity Index drug composite score.
Alcohol Use | 3 months after randomization and 6 months after randomization
  Frequency of alcohol use in past 30 days Revised Risk Behavior Assessment and breath test. Self-Report verified by biological sample Poisson.
  Addiction Severity Index alcohol composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Irma Kirtadze, MD, Principal Investigator — Addiction Research Center, Union Alternative Georgia, Tbilisi; Hendree Jones, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- Addiction Research Center, Union Alternative Georgia office, Tbilisi, Georgia

REFERENCES:
- [Background] Costenbader EC, Otiashvili D, Meyer W, Zule WA, Orr A, Kirtadze I. Secrecy and risk among MSM in Tbilisi, Georgia. AIDS Care. 2009 May;21(5):591-7. doi: 10.1080/09540120802385587. PMID 19444667
- [Background] Jones HE, Wong CJ, Tuten M, Stitzer ML. Reinforcement-based therapy: 12-month evaluation of an outpatient drug-free treatment for heroin abusers. Drug Alcohol Depend. 2005 Aug 1;79(2):119-28. doi: 10.1016/j.drugalcdep.2005.01.006. Epub 2005 Feb 24. PMID 16002021
- [Derived] Jones HE, Kirtadze I, Otiashvili D, Murphy K, O'Grady KE, Zule W, Krupitsky E, Wechsberg WM. Feasibility and initial efficacy of a culturally sensitive women-centered substance use intervention in Georgia: Sex risk outcomes. Subst Abuse Treat Prev Policy. 2015 Dec 8;10:47. doi: 10.1186/s13011-015-0043-0. PMID 26644132
- See also: Related Info — http://www.informaworld.com/smpp/title~content=t713403300